CLINICAL TRIAL: NCT04221932
Title: Implementation of Continuous Renal Replacement Therapy (CRRT) Key Performance Indicator (KPI) Reports to Standardize and Improve the Quality of CRRT Delivery in Alberta - "QUALITY-CRRT"
Brief Title: Implementation of CRRT KPI Reports to Standardize and Improve the Quality of CRRT Delivery in Alberta "QUALITY CRRT"
Acronym: QUALITY-CRRT
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Collaborators: Institute of Health Economics, Canada (Other); Alberta Innovates Health Solutions (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00075274
Record Dates: First submitted 2020-01-06; First posted 2020-01-09 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Critical Illness; Acute Kidney Failure
Keywords: Intensive Care Unit; Critical Illness; Acute Kidney Injury; Continuous Renal Replacement Therapy; Quality Improvement
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Pre Intervention: Retrospective evaluation of data from 2 years prior to the implementation of our CRRT KPI reports. This will include approximately 1500 participants.
  Interventions: Device: CRRT KPI Reports
- Post Intervention: This will be a prospective evaluation of all new ICU patients receiving CRRT in Alberta over a 2 year periods. This will include approximately 1500 participants
  Interventions: Device: CRRT KPI Reports

INTERVENTIONS:
Device: CRRT KPI Reports — This will involve the regular report of CRRT KPI reports across the CRRT programs across the province. It will also include standardization of CRRT practices across Alberta. Reports will include those for the program (i.e., structure), device (i.e., process) and patient outcomes (i.e., outcomes).

SUMMARY:
Acute kidney replacement therapy (i.e., dialysis) is used in 6-10% of patients admitted to intensive care units (ICUs). The amount of acute kidney replacement therapy use has increased in Canadian ICUs over the last several years. Continuous renal replacement therapy (CRRT) remains the most common form of acute renal replacement therapy used in ICUs.

Many different parts aspects of CRRT lack a usual way to be done, and because of this, are done differently in different ICUs. Not having generally accepted markers of the performance and delivery of CRRT is a main reason that we have these practice difference. This is an important gap in the way that clinicians deliver this important ICU therapy and is a main focus of ongoing research in ICU and dialysis.

The proposed project is a continuation of a program of work that first reviewed the current state of the quality and safety in ICU and dialysis. Then, a systematic review of all potential quality markers was done to see what options for measures were possible. Next, following a meeting of leaders of dialysis in the ICU, the most important of these measures were ranked to decide which ones could be used in monitoring CRRT for patients.

DETAILED DESCRIPTION:
Background: Renal replacement therapy (RRT) is a core life support technology used in approximately 1 in 10 ICU patients. RRT can be delivered intermittently or continuously. While intermittent RRT (IRRT) is used selectively in ICU settings, continuous RRT (CRRT) is the dominant initial form used worldwide. CRRT is a continuous method of blood purification that provides slow uninterrupted clearance of uremic toxins and enables acid-base, electrolyte and volume homeostasis while preserving hemodynamic stability. The, "Implementation of Continuous Renal Replacement Therapy (CRRT) Key Performance Indicator (KPI) Reports to Standardize and Improve the Quality of CRRT Delivery in Alberta - QUALITY-CRRT," is a proposed program of research to standardize and change the practice of CRRT in Alberta in order to improve the performance and delivery of this therapy to our most severely critically ill patients.

Last year in Alberta, 55.2% of patients were started on CRRT as an initial form of RRT. Patients receiving CRRT have greater illness severity (mean APACHE II score of 30.4 vs. 18.9), they are more likely to die (mortality of 41.3% vs. 7.3%) and have significantly increased healthcare utilization when compared to their non-CRRT receiving critically ill counterparts. In 2018, Alberta Health Services spent $2,437,097 to operate its CRRT program. However, these costs only include expendable supplies (i.e., fluids, filters, etc.) and do not include program maintenance or machine hardware expenses, thus underrepresenting the true cost of this therapy. In the setting of increasingly constrained healthcare resources, intervention is needed which may eliminate inefficiencies, improve performance, and decrease waste while ameliorating provider satisfaction and achieving better patient outcomes. Currently, clinicians do not routinely measure the performance of CRRT in Alberta (or elsewhere for that matter), and as such, are not in a position to understand or identify the inefficiencies or gaps in the quality of care of CRRT provided to critically ill patients.

The performance of CRRT may be measured by monitoring key performance indicators (KPIs). KPIs are necessary and can facilitate improved reliability of care, homogenize complex interventions, and provide a platform to measure and monitor performance and the impact of practice changes, and compliance with evidence-based standards. KPIs can be further used as targets for continuous quality improvement initiatives aimed at evaluating new or revised care processes, implementing new protocols or interventions, reducing variability in the delivery of healthcare and stimulating innovative research. The lack of validated and routinely reported KPIs for CRRT, however, are viewed as an important knowledge-to-care gap and may be associated with greater risk for suboptimal quality of CRRT delivery, and has been identified as a research priority.

To date, no Canadian program that has aimed to implement KPIs of CRRT care and to safeguard patients with the high-quality delivery of this complex technology. A focused program aimed to implement an inventory of KPIs for CRRT in order change practice and standardize care across a healthcare system to align with evidence-based best practices has the potential to transform the delivery of CRRT to critically ill patients. The proposed program of research will build upon previous phases of work that have identified and prioritized KPIs for CRRT care in order to implement these CRRT KPIs to change practice to provide effective, validated and standardized CRRT and ultimately to improve the quality of care to critically ill patients receiving CRRT by changing practice in order to decrease variation between all provincial CRRT programs so as to align with evidence-based CRRT best practices guidelines, therapies and prescriptions.

The Proposed Trial: QUALITY CRRT is an innovative, population-level, interrupted time series aimed to evaluate the effectiveness, safety and cost of implementing a multi-faceted CRRT quality assurance and improvement program in ICU settings. It will further explore the reach of QUALITY CRRT by extending the ongoing work on public and patient/family understanding of participation in low-risk ICU research trials focused on generating and implementing best practices. This work will provide insights into the perceived value of such research for Canada's healthcare system as well as to demonstrate feasibility, to build capacity for future population-level pragmatic trials focused on health systems innovations and quality improvement/assurance in ICU settings, and to continue to engage the public in the healthcare and critical care research processes.

Prior to the implementation of the CRRT quality assurance and improvement program and reporting of CRRT KPIs, each ICU will have a minimum 24 months of baseline data analyzed followed by 24 months of prospective data. Long-term outcomes (i.e., individual and healthcare systems costs) will be determined through a future outcome modelling process. During the entire study period participants will be included into the study. Prior to the reporting of CRRT KPIs, there will be provincial and site educational events to prepare local experts, champions and educators in preparation for implementation of CRRT KPI reporting. These reports will be available at each site to their respective healthcare professionals, local champions, as well as to the study Executive, Steering and Quality Monitoring Committees. Following the implementation of CRRT KPI reporting, the study team will review the CRRT KPI reports at each site on a quarterly basis and will relay these results to individual unit stakeholders and champions. Any educational events of quality initiatives will be led by individual units but will be recorded as a treatment outcome.

QUALITY CRRT will compare a novel approach to monitoring the delivery of CRRT to critically ill patients. For the study intervention, a multi-faceted CRRT quality assurance and improvement program will be implemented to CRRT programs across Alberta. This will include a review of the individual unit CRRT KPI reports, followed by in person as well as tele/video targeted information sessions led by members of our steering committee. Reports will also be provided for each unit that will be distributed to all CRRT providers and stakeholders. The current practice of CRRT will be determined by interrogating our CIS for 24 months preceding our study intervention to determine baseline CRRT performance. This will frame the counterfactual scenario for the interrupted-time series analysis.

In the usual care (i.e., current practice), CRRT will be monitored as per unit-specific parameters. For the study intervention, each CRRT program will be ensured to have appropriate leadership and education (i.e., structure KPIs) in place. CRRT KPI reporting (i.e., quarterly reports for filter life, downtime, delivered dose, access alarms, adverse events and ICU mortality) will be implemented and reviewed at both a trial, and unit specific level performed ad hoc and at quarterly intervals. During the systems level implementation of CRRT KPIs, each ICU will receive a multi-faceted education tailored to each ICU and informed by local CRRT leaders. The evidence-based multi-faceted strategy will maximize the utilization of the CRRT KPI reports. Our implementation strategy will include, 1) inter-professional educational strategies (grand rounds, seminars, webinars), 2) site champions, 3) quarterly audit and feedback reports and 4) quarterly tele/videoconference and in-person visits. While the strategy will contain similar themes at each site, individual components will be customized in order to address unit specific shortcomings in their CRRT KPI performance. Each site will be encouraged to facilitate and conduct their own audit and educational activities. A central website repository of typical troubleshooting tools for high-yield interventions on KPIs not achieving our proposed benchmarks will be developed and available for reference.

QUALITY CRRT will enroll all new ICU admissions receiving CRRT in the 13 adult and 2 pediatric ICUs in Alberta who provide this therapy. In 2018 there were 12,132 adult and 1,592 pediatric admission per year with 5.6% and 1.4% of these patients (i.e., 680 adult and 22 pediatric patients) receiving CRRT in these 15 ICUs. We are planning to conduct this study over a 2-year period, for a total of approximately 1,500 adult and pediatric participants, over nearly 25,000 patient-days. As all patient data can be retrieved from our CIS, it is anticipated that the loss to follow up to be minimal.

Data will be compiled retrospectively prior to the reporting of CRRT KPIs and implementation of the multi-faceted quality assurance and improvement program; after data will be collected following this implementation. Analysis will be conducted between the pre- and post-implementation groups. Analyses of the primary and secondary outcomes will involve summary measures obtained by aggregating the endpoints. Analyses will be performed using the Stata software package (StataCorp, Texas, USA). Baseline comparisons will be performed using chi-squared test for equal proportions with results to be reported as numbers, percentages, and 95% confidence intervals. Continuous normally distributed variables will be compared using paired t-tests and reported as means with 95% confidence intervals, while non-normally distributed will be compared using Wilcoxon rank sum tests and reported as medians and interquartile ranges (IQRs). In case of small sample size, fisher's exact test will be used. Descriptive and multivariable analysis will be performed to adjust for important risk factors and to understand the difference between variables.

Pre-specified subgroup analysis will include ICU patients to 1) adult vs. pediatric, 2) female vs. male, 3) academic vs. community ICUs, 4) cardiovascular ICUs vs. medical/surgical ICUs, 5) high volume vs. low volume centers (i.e., as per quartiles). We will perform the above analyses for health economic evaluations, patient and process of case measures to include our pre-specified primary and secondary outcomes for each subgroup. Each analysis will be accompanied by a test for interaction between treatment and subgroup to ascertain whether effects differ significantly between subgroups.

Trial Management: The data coordinating and management centre is the Institute of Health Economics (IHE) in Edmonton, Alberta. The IHE will be responsible for data management, analysis, progress updates and for developing site-specific quarterly CRRT Quality Dashboard reports. The IHE will liaise with study committees, individual site champions and applicable partners. The QUALITY CRRT study will have an Executive Committee Responsible to overall trial management. There will also be a Steering Committee with stakeholders from each site to review the quarterly reports. Finally, QUALITY CRRT will have an international Quality Monitoring Committee that the Executive Committee will liaise with the ensure appropriate trial oversight.

Significance, Capacity Building and Impact: QUALITY CRRT will serve to implement an evidence-based CRRT Quality Dashboard. The findings of QUALITY CRRT will underscore the importance and need to widely implement a CRRT Quality Dashboard, not just in Alberta, but in any healthcare system which provides CRRT.

ELIGIBILITY:
Inclusion Criteria:

* ICU admission
* CRRT initiation

Exclusion Criteria:

- None

Min Age: 1 Year | Sex: All
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — It is imperative that sex and gender be considering and explored in any health services program. Gender identification will not be captured in this work. However, sex will be evaluated in QUALITY CRRT. QUALITY CRRT will include all patients, both men and women, receiving CRRT in adult ICUs in Alberta in an unbiased fashion through our current and future CISs, eCritical and ConnectCare™, respectively. Our analyses will be stratified by sex to explore if there is a difference in CRRT treatment and quality by sex. Further, it is recognized that there is a biological sex and gender identity gap in health research. To help address this gap, we will ensure that 50% of all research executive, steering committee and quality monitoring committee members are women. QUALITY CRRT will also consider sex/gender in the planning, conduct and dissemination of all aspects of QUALITY CRRT.
Study Population: All Alberta critically ill patients requiring CRRT.
Sampling Method: Non-Probability Sample
Enrollment: 945 (Actual)
Dates: Start 2022-07-05 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Quality of CRRT performance and delivery | 2 years post intervention
  Quarterly changes in the performance of the CRRT KPIs following the initiation of CRRT KPI reporting and our multi-faceted quality assurance and improvement knowledge translational intervention. The specific CRRT KPIs will include, but will not necessarily be limited to, 1) CRRT leadership; 2) CRRT education; 3) average filter life measured in hours; 4) downtime in percentage of treatment time lost; 5) average dose prescribed and delivered in ml/kg/hr; 6) alarms in number/day/machine; 7) significant adverse events as per number of reporting & learning system (RLS) records/month; and 8) ICU mortality. Based on the vanguard phase there may be additional or further refined KPIs to consider. These outcomes will be recorded on a continual quarterly basis to determine the predicted slope change impact following the implementation of our intervention.

SECONDARY OUTCOMES:
Economic Evaluation | 3 years post intervention
  The economic evaluation will comprise two parts: 1) a within-study analysis, and 2) a longer term, model based, analysis. The within-study analysis will focus on costs and outcomes collected during the study period. The longer-term model-based analysis will supplement the study data with data from literature, particularly patient outcomes. The additional data will be used to estimate the cost-effectiveness of QUALITY CRRT when longer terms outcomes are taken into consideration. The within-study evaluation will focus on CRRT costs. It will include total quarterly unit-specific CRRT-associated costs following the implementation of the CRRT KPI reporting program. It will also determine healthcare systems costs to include total ICU and hospital stay associated costs, ongoing new end-stage renal disease (i.e., chronic RRT) costs, total healthcare costs, patient life-years gained and quality-adjusted life years (QALY).
Patient-centred Outcomes | 3 years post intervention
  This will include ICU, hospital and 90-day mortalities, ICU and hospital lengths of stay, duration of CRRT and IRRT treatment, and renal recovery measured at 6 months. While this study is not designed to evaluate the effect that the implementation of the reporting of CRRT KPIs will have on mortality, lengths of treatment and stay or renal recovery, these are important patient-centered outcomes that will need to be considered as balancing measures for CRRT KPI reporting and implementation of the multi-faceted knowledge translation intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Oleksa G Rewa, MD MSc, Principal Investigator — University of Alberta
Locations (14):
- Canada (14):
  - Alberta Children's Hospital, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - Rockyview General Hospital, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - Stollery Childrens Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Red Deer Regional Hospital, Red Deer, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta
  - Grey Nuns Community Hospital, Edmonton, Albert
  - Mazankowski Alberta Heart Institute, Edmonton, Albert

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Opgenorth D, Reil E, Lau V, Fraser N, Zuege D, Wang X, Bagshaw SM, Rewa O. Improving the quality of the performance and delivery of continuous renal replacement therapy (CRRT) to critically ill patients across a healthcare system: QUALITY CRRT: a study protocol. BMJ Open. 2022 Feb 4;12(2):e054583. doi: 10.1136/bmjopen-2021-054583. PMID 35121604